CLINICAL TRIAL: NCT00986765
Title: Low Molecular Weight Heparin, Enoxaparin, to Prevent Adverse Maternal and Perinatal Outcomes in Women With Previous Severe Preeclampsia at Less Than 34 Weeks' Gestation. A Prospective Randomized Trial
Brief Title: Prevention of Maternal and Perinatal Complications by Enoxaparin in Women With Previous Severe Preeclampsia
Acronym: HEPEPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P071211
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Preeclampsia
Keywords: Fetal growth restriction; Abruptio placentae; Perinatal death
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Abruptio Placentae; Perinatal Death | interventions — Enoxaparin; acetylsalicylic acid lysinate; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovenox® , 4000 UI/day (+ Aspegic®) (Experimental): Lovenox® (enoxaparin), 4000 UI/day (+ Aspegic® (Aspirin), 100 mg)
  Interventions: Drug: Lovenox® (enoxaparin)
- Aspegic ®, 100 mg/day (Active Comparator): Aspegic® (Aspirin),100 mg/day
  Interventions: Drug: Aspegic ® (Aspirin)

INTERVENTIONS:
Drug: Lovenox® (enoxaparin) — Injectable solution 4000 UI
  Arms: Lovenox® , 4000 UI/day (+ Aspegic®)
Drug: Aspegic ® (Aspirin) — 100 mg/day
  Arms: Aspegic ®, 100 mg/day

SUMMARY:
Preeclampsia (PE) complicates 2-8% of pregnancies. It is associated with an increased risk of adverse maternal (death, eclampsia, abruptio placenta, HELLP syndrome) and perinatal (perinatal death, growth restriction, prematurity) outcomes. The only definite treatment of PE remains pregnancy termination. Therefore, prevention of PE remains an important challenge. Low dose aspirin may be used in the prevention of PE, particularly in women who had a severe preeclampsia before 34 weeks. Its efficiency, however, is very weak. Recently, it has been suggested that low molecular weight heparin might be useful in the prevention of PE.

The aim of this study is to analyze the usefulness of the enoxaparin 4000 UI/day in the prevention of a composite maternal or perinatal morbidity (occurrence of one of the following events: maternal death, PE, fetal growth retardation, abruptio placenta, perinatal death) in women who previously had a severe preeclampsia at less than 34 weeks' gestation. To answer this question, the investigators propose to conduct a multicenter prospective randomized trial that will compare two groups in parallel: a group where women will have an association of enoxaparin 4000 U/day and aspirin 100 mg/day and another group where women would have only aspirin 100 mg/day. The number of patients needed is 255 (amendment n°2-approved 06/12/2011) .

DETAILED DESCRIPTION:
1. Purpose of the study: To determine whether low molecular weight heparin (LMWH) enoxaparin decreases the rate of maternal and perinatal composite morbidity in women who previously had a severe preeclampsia that occurred at less than 34 weeks' gestation.
2. Patients and methods: Multicenter, prospective, randomized trial comparing 2 groups of patients:

   * First group treated with aspirin 100 mg/day until 35 weeks' gestation and enoxaparin subcutaneous 4000 UI/day until delivery.
   * Second group treated with aspirin 100 mg/day alone until 35 weeks' gestation.

   At first prenatal visit between 7-13 weeks, inclusion and exclusion criteria will be searched. Randomization will be performed by internet software. It will be performed by center.

   After randomization at first prenatal visit patients will be allocated to aspirin-enoxaparin or aspirin alone as mentioned above. Enoxaparin will be stopped the day of delivery or after the occurrence of a complication that necessitates delivery. Pregnancy management will be performed as recommended by standard care. Each month, blood samples will be drawn for platelets count and the analysis of angiogenic factors (sFlt1, sEng, free PlGF and VEGF). In addition, blood sample will be drawn at first prenatal visit for thrombophilia work-up (Prot C, Factor V Leiden, Prothrombin gene polymorphism). Only results of platelet count will be given to local investigators during the study. All other analysis will be performed at the end of the study by Pr Gris at NIMES, and will be blinded to clinical results.
3. Statistical analysis: Women with previous severe preeclampsia at less than 34 weeks' gestation have a 40% risk of occurrence of a composite morbidity (primary outcome defined above) at the next pregnancy. A 33% decrease of the composite morbidity defined above in women treated with LMWH enoxaparin is considered to be efficient. With an alpha risk of .05 and a beta risk of .20, the number of patients needed is 255 (amendment n°2-approved 06/12/2011) . This trial will be analyzed as an "Intention to treat study". No interim analysis for the primary outcome will be performed. Results will be stratified by center.

   Primary outcome (categorical variable) will be analyzed by chi-square test. Secondary outcomes will analyzed by chi-square test for categorical variables or ANOVA for continuous variables.

   Statistical significance will be considered with a p value <.05. Statistical analysis will be performed by STATA software (StataCorp, 2003, TX).
4. Registry of non-included patients: Each patient that has been non-eligible for the trial will be noted in a registry as well as the reason of exclusion.
5. Independent committee for analysis of adverse outcome: An independent committee will analyze adverse maternal and perinatal outcomes before statistical analysis at the end of the study. This analysis will be blinded for the treatment allocated for the patients.
6. Definitions:

   * Preeclampsia: Preeclampsia is defined by the association of gestational hypertension (after 20 weeks' gestation, a systolic blood pressure > 140 mmHg and/or a diastolic blood pressure > 90 mmHg, persistent at least at 4 hours apart, or a persistent diastolic blood pressure > 110 mmHg) and proteinuria (24 hours proteinuria > 300 mg, or at least 1+ persistent at least at 4 hours apart).
   * Fetal growth restriction: Fetal growth restriction is defined by a birthweight < 10th percentile.
   * Abruptio placentae: Abruptio placenta is defined by the association of bleeding and one of the following criteria:

     * Abnormal fetal heart rate,
     * Abdominal pain,
   * Perinatal death: Perinatal death is a death that occurs during fetal or neonatal Period, from 22 weeks' gestation until the 28th day of life.
   * Severe preeclampsia is defined, in a woman with preeclampsia, by the presence of one of the following criteria:

Maternal:

* Severe hypertension (systolic blood pressure >160 MmHg and/or diastolic blood pressure > 110 mm Hg),
* Persistent headaches or visual disturbances,
* Persistent epigastric or RUQ pain,
* 24 hours proteinuria ≥ 5gr,
* Oliguria < 500 ml/24h, or serum creatinine > 120 µmol/L,
* Eclampsia,
* Pulmonary edema,
* Abruption,
* Platelet count < 100,000/ µL,
* lactate dehydrogenase (LDH) > 600U/L, aspartate transaminase (ASAT) > 2 normal.

Fetal:

* Severe fetal growth restriction (< 5ème percentile)
* Severe Oligohydramnios.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Patient with a previous severe preeclampsia that occurred at less than 34 weeks' gestation
* Patient between 7 and 13 weeks +6 days at first prenatal visit
* Singleton pregnancy
* Affiliation to social security
* Informed consent given after receiving information on the study.

Exclusion Criteria:

* Patient under law protection
* Inability to sign written consent
* Inability to follow the protocol because of a psychiatric disease
* History of deep venous thromboembolism during previous pregnancy
* Need of low molecular weight heparin during pregnancy
* Previous arterial thrombosis
* Patient having a cardiac valvular prosthesis that necessitates anticoagulation during pregnancy
* Renal failure (creatinine clearance < 30 ml/min, or serum creatinine > 180 µmol/L
* Previous hemorrhagic disease
* A disease that might bleed (gastric ulcer)
* Antiphospholipid antibody syndrome
* Allergy to Aspirin
* Allergy to heparins
* Thrombocytopenia related to heparin use
* Thrombocytopenia <100,000 /µL at first prenatal visit
* Antecedent of osteoporosis
* Inability to do subcutaneous injection of heparin
* Weight > 100 kg
* Patient included in another interventional trial
* Patient positive for anti-phospholipids antibodies
* Patient positive for HIV or HCV or HBS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2009-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a composite morbidity that may occur : maternal death, or perinatal death, or preeclampsia, or abruptio placenta, or fetal growth restriction. | from randomization until one month after the delivery

SECONDARY OUTCOMES:
Recurrence of preeclampsia alone | from randomization until one month after the delivery
Recurrence of severe preeclampsia | from randomization until one month after the delivery
Fetal growth restriction alone | from randomization until one month after the delivery
Severe fetal growth restriction (< 5th percentile) | from randomization until one month after the delivery
Perinatal death alone | from randomization until one month after the delivery
Neonatal death | from randomization until one month after the delivery
Abruption alone | from randomization until one month after the delivery
Maternal death | from randomization until one month after the delivery
Fetal loss (10-21 weeks) | from randomization until one month after the delivery
Fetal death | from 15 weeks to delivery
Recurrence of preeclampsia controlled for thrombophilia analysis (polymorphism of factor V Leiden, prothrombin G20210A gene polymorphism) | from randomization until one month after the delivery
Recurrence of preeclampsia controlled for angiogenic factors (free VEGF and PlGF, sFlt1, sEng) | from randomization until one month after the delivery
Neonatal morbidity (NICU transfer, length of hospitalization, mechanical ventilation > 24 hours, respiratory distress syndrome, necrotizing enterocolitis, periventricular leucomalacia, bronchopulmonary dysplasia, intraventricular hemorrhage grade III-IV) | from randomization until one month after the delivery
Enoxaparin toxicity: hemorrhage, skin reaction, thrombocytopenia (<100000/µL) related to heparin | from randomization until one month after the delivery
Bone fracture | from randomization until one month after the delivery

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Haddad, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

REFERENCES:
- [Derived] Lecarpentier E, Gris JC, Cochery-Nouvellon E, Mercier E, Abbas H, Thadhani R, Karumanchi SA, Haddad B. Urinary Placental Growth Factor for Prediction of Placental Adverse Outcomes in High-Risk Pregnancies. Obstet Gynecol. 2019 Dec;134(6):1326-1332. doi: 10.1097/AOG.0000000000003547. PMID 31764746
- [Derived] Lecarpentier E, Gris JC, Cochery-Nouvellon E, Mercier E, Touboul C, Thadhani R, Karumanchi SA, Haddad B. Angiogenic Factor Profiles in Pregnant Women With a History of Early-Onset Severe Preeclampsia Receiving Low-Molecular-Weight Heparin Prophylaxis. Obstet Gynecol. 2018 Jan;131(1):63-69. doi: 10.1097/AOG.0000000000002380. PMID 29215518
- [Derived] Haddad B, Winer N, Chitrit Y, Houfflin-Debarge V, Chauleur C, Bages K, Tsatsaris V, Benachi A, Bretelle F, Gris JC, Bastuji-Garin S; Heparin-Preeclampsia (HEPEPE) Trial Investigators. Enoxaparin and Aspirin Compared With Aspirin Alone to Prevent Placenta-Mediated Pregnancy Complications: A Randomized Controlled Trial. Obstet Gynecol. 2016 Nov;128(5):1053-1063. doi: 10.1097/AOG.0000000000001673. PMID 27741174